CLINICAL TRIAL: NCT02533232
Title: Minocycline Augmentation of Clozapine for Treatment Resistant Schizophrenia: A Randomised Placebo-controlled Double-blind Trial
Brief Title: Minocycline Augmentation of Clozapine for Treatment Resistant Schizophrenia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PILL-MAC-001
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Anti-inflammatory; Clozapine; Minocycline; Psychosis NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; cyclopia sequence; Mental Disorders | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Matching placebo for Minocycline
  Interventions: Drug: Minocycline
- Minocycline (Experimental): Minocycline 200mg once a day orally
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 200mg per day
  Other Names: Mesodrum

SUMMARY:
This a randomized double-blind placebo controlled trial which aims to determine the beneficial effects of minocycline augmentation to clozapine in partial responders to Treatment Resistant Schizophrenia (TRS).

DETAILED DESCRIPTION:
The primary objective is to determine if the addition of minocycline to Clozapine, Treatment as Usual (TAU) Improves negative symptoms and/or positive symptoms.

The secondary objectives are to determine:

* Effects on cognitive functioning.
* Effects on social functioning and quality of life.
* Safety and tolerability.
* Possible additive effects of Minocycline added to TAU
* The effect on inflammatory biomarkers associated with schizophrenia. Both pro and anti-inflammatory cytokines will be drawn at baseline and endpoint. We will test to see if minocycline is associated with improvements in abnormal cytokines as compared to placebo.

The study will be a randomized double-blind placebo controlled trial of minocycline added to clozapine (Treatment as Usual) in TRS. There will be two treatment arms: one arm receiving TAU with minocycline and the other TAU with placebo for a period of twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 18-65 years, IQ >70 (to complete assessments) identified by treating psychiatrist.
* Confirmation of schizophrenia by using The MINI psychiatric interview (at baseline only)
* Assessed as competent to provide informed consent by treating psychiatrist.
* Antipsychotic medication has remained stable 4 weeks prior to baseline *. Assessed as a partial responder to clozapine: patients prescribed clozapine at a stable therapeutic dose for a minimum of 3 months with total Positive and Negative Syndrome Schizophrenia (PANSS) score >70.

Exclusion Criteria:

* Prior history of intolerance or serious side effects (hepatotoxicity, photosensitivity, blood dyscrasias) to any of the Tetracyclines.
* Concomitant Penicillin therapy or concomitant anticoagulant therapy.
* Active substance abuse (except nicotine or caffeine) or dependence within the last three months according to ICD 10 criteria.
* Treatment with Warfarin or Lamotrigine.
* Current or previous treatment with minocycline or other tetracycline antibiotics in the preceding three months before study entry.
* Relevant current or past hematologic, hepatic, renal, neurological or other medical disorder that in the opinion of the principal investigator may interfere with the study.
* Pregnant or breast-feeding females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale PANSS | 3 months
  PANSS is an assessment measures to assess severity of symptoms of schizophrenia

SECONDARY OUTCOMES:
CogState | 3 Month
  Measuring all seven domains recommended by MATRICS (NIMH initiative). These domains include speed processing, attention/vigilance, Working memory (nonverbal & verbal), verbal learning, visual learning, reasoning and problem solving and social cognition's.

OTHER OUTCOMES:
Social Functioning Scale | 3 Month
  Self-rating questionnaire assessing social functioning in 7 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Inti Qurashi, MD, Principal Investigator — Manchester University ,UK
Locations (4):
- Pakistan (4):
  - Abasi Shaheed Hospital, Karachi, Sindh
  - Civil hospital Karachi, Karachi, Sindh
  - Karwn e Hayat, Karachi, Sindh
  - Institute of Behavioral Sciences, Karachi, Sindh

REFERENCES:
- [Background] Qurashi I, Collins JD, Chaudhry IB, Husain N. Promising use of minocycline augmentation with clozapine in treatment-resistant schizophrenia. J Psychopharmacol. 2014 Jul;28(7):707-8. doi: 10.1177/0269881114527358. Epub 2014 Mar 19. PMID 24646811
- [Background] Conley RR, Buchanan RW. Evaluation of treatment-resistant schizophrenia. Schizophr Bull. 1997;23(4):663-74. doi: 10.1093/schbul/23.4.663. PMID 9366002
- [Background] Chakos M, Lieberman J, Hoffman E, Bradford D, Sheitman B. Effectiveness of second-generation antipsychotics in patients with treatment-resistant schizophrenia: a review and meta-analysis of randomized trials. Am J Psychiatry. 2001 Apr;158(4):518-26. doi: 10.1176/appi.ajp.158.4.518. PMID 11282684
- [Background] Rossler W, Salize HJ, van Os J, Riecher-Rossler A. Size of burden of schizophrenia and psychotic disorders. Eur Neuropsychopharmacol. 2005 Aug;15(4):399-409. doi: 10.1016/j.euroneuro.2005.04.009. PMID 15925493
- [Background] Sommer IE, Begemann MJ, Temmerman A, Leucht S. Pharmacological augmentation strategies for schizophrenia patients with insufficient response to clozapine: a quantitative literature review. Schizophr Bull. 2012 Sep;38(5):1003-11. doi: 10.1093/schbul/sbr004. Epub 2011 Mar 21. PMID 21422107
- [Background] Lin A, Kenis G, Bignotti S, Tura GJ, De Jong R, Bosmans E, Pioli R, Altamura C, Scharpe S, Maes M. The inflammatory response system in treatment-resistant schizophrenia: increased serum interleukin-6. Schizophr Res. 1998 Jun 22;32(1):9-15. doi: 10.1016/s0920-9964(98)00034-6. PMID 9690329
- [Background] van Berckel BN, Bossong MG, Boellaard R, Kloet R, Schuitemaker A, Caspers E, Luurtsema G, Windhorst AD, Cahn W, Lammertsma AA, Kahn RS. Microglia activation in recent-onset schizophrenia: a quantitative (R)-[11C]PK11195 positron emission tomography study. Biol Psychiatry. 2008 Nov 1;64(9):820-2. doi: 10.1016/j.biopsych.2008.04.025. Epub 2008 Jun 4. PMID 18534557
- [Background] Farber NB. The NMDA receptor hypofunction model of psychosis. Ann N Y Acad Sci. 2003 Nov;1003:119-30. doi: 10.1196/annals.1300.008. PMID 14684440
- [Background] Javitt DC, Zukin SR. Recent advances in the phencyclidine model of schizophrenia. Am J Psychiatry. 1991 Oct;148(10):1301-8. doi: 10.1176/ajp.148.10.1301. PMID 1654746
- [Background] Labrie V, Roder JC. The involvement of the NMDA receptor D-serine/glycine site in the pathophysiology and treatment of schizophrenia. Neurosci Biobehav Rev. 2010 Mar;34(3):351-72. doi: 10.1016/j.neubiorev.2009.08.002. Epub 2009 Aug 18. PMID 19695284
- [Background] Anticevic A, Gancsos M, Murray JD, Repovs G, Driesen NR, Ennis DJ, Niciu MJ, Morgan PT, Surti TS, Bloch MH, Ramani R, Smith MA, Wang XJ, Krystal JH, Corlett PR. NMDA receptor function in large-scale anticorrelated neural systems with implications for cognition and schizophrenia. Proc Natl Acad Sci U S A. 2012 Oct 9;109(41):16720-5. doi: 10.1073/pnas.1208494109. Epub 2012 Sep 25. PMID 23012427
- [Background] Deakin JF, Lees J, McKie S, Hallak JE, Williams SR, Dursun SM. Glutamate and the neural basis of the subjective effects of ketamine: a pharmaco-magnetic resonance imaging study. Arch Gen Psychiatry. 2008 Feb;65(2):154-64. doi: 10.1001/archgenpsychiatry.2007.37. PMID 18250253
- [Background] Meltzer HY. Treatment-resistant schizophrenia--the role of clozapine. Curr Med Res Opin. 1997;14(1):1-20. doi: 10.1185/03007999709113338. PMID 9524789
- [Background] Domercq M, Matute C. Neuroprotection by tetracyclines. Trends Pharmacol Sci. 2004 Dec;25(12):609-12. doi: 10.1016/j.tips.2004.10.001. PMID 15530637
- [Background] Tikka T, Fiebich BL, Goldsteins G, Keinanen R, Koistinaho J. Minocycline, a tetracycline derivative, is neuroprotective against excitotoxicity by inhibiting activation and proliferation of microglia. J Neurosci. 2001 Apr 15;21(8):2580-8. doi: 10.1523/JNEUROSCI.21-08-02580.2001. PMID 11306611
- See also: Website of Pakistan Institute of Learning and Living — http://pill.org.pk